CLINICAL TRIAL: NCT05595746
Title: Evaluation of the Relationship Between Vertical Mucosal Thickness and Radiological Bone Loss of Platform-Switching Implants Placed at Different Levels
Brief Title: Radiological Bone Loss on Different Levels of Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berceste Guler, Assoc. Prof., Kutahya Health Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-05/07
Record Dates: First submitted 2022-10-16; First posted 2022-10-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Alveolar Bone Loss; Peri-Implantitis; Bone Loss in Jaw
Keywords: vertical mucosal height; dental implant; marginal bone loss; keratinized gingival width
MeSH Terms: conditions — Alveolar Bone Loss; Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Controlled, non-randomized, single-blind, parallel
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are assigned a number by hiding their names. While the measurements are being made, the researcher does not know which group the participant belongs to. All radiographic and clinic measurements are collected in one file.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- equicrestally placement with higher vertical mucosa (Experimental): Implants with a vertical mucosal height greater than 2 mm (A) and placed equicrestally (I) are in group A-I.
  Interventions: Procedure: dental implant placement
- subcrestally placement with higher vertical mucosa (Experimental): Implants with a vertical mucosal height greater than 2 mm (A) and placed subcrestally (II) are in group A-II.
  Interventions: Procedure: dental implant placement
- equicrestally placement with less vertical mucosa (Experimental): Implants with a vertical mucosal height of 2 mm or less (B) and placed equicrestally (I) are in group B-I.
  Interventions: Procedure: dental implant placement
- subcrestally placement with less vertical mucosa (Experimental): Implants with a vertical mucosal height of 2 mm or less (B) and placed subcrestally (II) are in group B-II.
  Interventions: Procedure: dental implant placement

INTERVENTIONS:
Procedure: dental implant placement — In dental implant placement surgery, first of all, intraoral infiltrative anesthesia is applied to the area. After the crestal incision, the buccal flap is elevated to full thickness. Vertical mucosal height is measured with a William type standard periodontal probe. The palatal/lingual flap is then elevated to full thickness. The implant is placed at different levels with the standard protocol determined by the manufacturer. Study groups are determined by the placement levels of the implants and the vertical mucosal height measurement values. After the implants are placed, the flap is closed primarily.

SUMMARY:
One of the criteria used for long-term implant success is the evaluation of radiographic bone loss. It is known that the keratinized mucosa over the alveolar crest forms a protective barrier against inflammatory infiltration. In addition, it has been reported that the vertical mucosal thickness on the crest is important in the formation of the biological width around the implant. The aim of this study was to evaluate the effect of vertical mucosal thickness on the alveolar crest on peri-implant marginal bone loss around crestal and subcrestal placed platform-switching implants. In this study, patients will be divided into 2 main groups with vertical mucosal thickness of 2 mm and less and more than 2 mm, and both groups will consist of 2 subgroups as crestally and subcrestally according to the implant level placed. A total of 80 implants will be included, 20 implants in each group. Before starting the surgery, after anesthesia is given, the width of the patient's peri-implant keratinized mucosa and the vertical mucosal thickness over the alveolar crest will be measured. Clinical and radiological measurements will be made in all patients during the prosthetic loading session (T0), at 3rd month (T1), 6th month (T2) and 1 year after loading (T3). With standardized control periapical radiographs to be taken as a result of one-year follow-up, the marginal bone loss amount in the implants will be evaluated using soft-ware.

DETAILED DESCRIPTION:
Dental implants have become one of the most common treatments used for the rehabilitation of lost teeth. The success rate of dental implant treatment is quite high. One of the criteria used for long-term implant success is the evaluation of radiographic bone loss. It is known that the keratinized mucosa over the alveolar crest forms a protective barrier against inflammatory infiltration. It has been reported that the vertical mucosal thickness over the alveolar crest in the operation area before dental implant treatment is important in the formation of the biological width around the implant. There are studies in the literature examining the effects of vertical mucosal thickness on peri-implant marginal bone loss. In a study presented by Linkevicius et al., in 2014, they divided 80 patients into 2 groups according to their mucosal thickness. It was reported that radiological bone loss was 1.17 mm in the group with low vertical mucosal thickness at the end of 1-year follow-up, and 0.21 mm in the group with high vertical thickness.

The aim of the study was to evaluate the effect of vertical mucosal thickness on the alveolar crest on peri-implant marginal bone loss around crestal and subcrestal placed platform-switching implants.

Before starting the surgery, after the patient is anesthetized, the width of the peri-implant keratinized mucosa and the vertical mucosal thickness over the alveolar crest will be measured. In this study, patients will be divided into 2 main groups with vertical mucosal thickness of 2 mm and less and more than 2 mm, and both groups will consist of 2 subgroups as crestal and subcrestal according to the implant level placed.

It is planned to use the same brand of implant and platform-switch abutment in patients. With standardized control periapical radiographs to be taken as a result of one-year follow-up, the marginal bone loss amount in the implants will be evaluated using software. Routine clinical and radiological measurements will be repeated in all patients at the prosthetic loading session (T0), at 3 months (T1), at 6 months (T2), and 1 year after loading (T3). Pre-surgical radiographs will be taken from the patients who participated in our study, as in all implant patients Clinical measurements.

1. Plaque index (Löe & Silness) and gingival index (Silness & Löe) are obtained by measuring 4 regions of a tooth (mesial, distal, buccal and lingual) with a Williams periodontal probe.

   Attachment loss: It is the value of the distance between a tooth and the free gingiva, based on the enamel-cementum junction, measured using a Williams periodontal probe.
2. Bleeding on probing index (Ainamo & Bay): In this index, probing is performed by gently walking around the pocket. As a result of probing, the evaluation is made by looking at the presence or absence of bleeding in the gingiva. A positive value is given if bleeding occurs within 10-15 seconds after probing in the mesial, distal, buccal and lingual gingival parts of all teeth. The ratio of the bleeding area to the examined area is expressed as %.
3. Keratinized gingival width: It is the distance from the free gingival margin to the mucogingival junction line.
4. Vertical mucosal thickness: It is the distance from the apex of the alveolar crest to the gingival margin. It will be measured with a standardized William type probe.
5. Pocket depth: The vertical distance between the base of the periodontal sulcus and the gingival margin with a standard periodontal probe.
6. Peri-implant pocket depth: It is the vertical distance between the base of the peri-implant sulcus and the gingival margin.
7. Marginal bone level: Radiographic evaluation of the distance between the restoration margin and the bone level.

Sample Selection: Taking the effect size of 0.08 for the significance value in the G Power analysis program as a reference to a previously presented study, 60 implants were planned to be taken for α= 0.05 and 80% power. However, since the study is a long-term control study, it is planned to take 20 implants each, due to the risk of patients not coming to the control sessions. A total of 80 implants will be included.

Statistical analysis method: All analyzes will be done with (Statistical Package for the Social Sciences) SPSS software. In-group temporal evaluations in test and control groups will be evaluated using Paired sample -T or Wilcoxon test according to normal distribution values. For comparisons between groups, the data will be analyzed by independent sample-T or Mann Whitney U test according to their normal distribution. The normal distribution of the data will be evaluated with the Kolmogorov-Smirnov test. The significance value will be taken as 0.05. Relationships between variables will be evaluated with Logistic Regression Analysis or Multivariate Regression Analysis.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* The patient does not have any systemic disease
* Implants are placed in the fully healed alveolar bone
* There is no need for horizontal and vertical augmentation in the area where the implant will be placed.
* Interocclusal distance higher than 7 mm
* Cooperative patients
* At least 9 mm of alveolar bone in the patient's mandible or maxilla in the area where the implant will be placed

Exclusion Criteria:

* Pregnant and lactation
* Mentally retarded patients
* Immediate loading
* Alveolar bone defects
* Smoking more than 10 cigarettes per a day
* Immunsupression or deficiency on bone metabolism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Radiographic peri-implant marginal bone loss | 1 year after prosthetic loading
  It is the result to be obtained by radiographic evaluation of peri-implant marginal bone loss of 4 study groups formed by vertical mucosal height and implant placement levels.

SECONDARY OUTCOMES:
Marginal bone loss related keratinized gingival height | 1 year after prosthetic loading
  Peri-implant marginal bone loss with keratinized gingival height
Marginal bone loss related keratinized gingival thickness | 1 year after prosthetic loading
  Peri-implant marginal bone loss with keratinized gingival thickness
Evaluation of clinical peri-implant health with plaque index | 1 year after prosthetic loading
  Peri-implant plaque index clinical data will be used.
Evaluation of clinical peri-implant health with gingival index | 1 year after prosthetic loading
  Peri-implant gingival index clinical data will be used.
Evaluation of clinical peri-implant health with bleeding on probing index | 1 year after prosthetic loading
  Peri-implant bleeding on probing clinical data will be used.
Evaluation of clinical peri-implant health with pocket depth on probing index | 1 year after prosthetic loading
  Peri-implant pocket depth on probing clinical data will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Güler, Study Director — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Department of Periodontology, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be shared if the principal investigator is contacted.
Supporting Information: Study Protocol, ICF
Time Frame: Following acceptance of manuscript
Access Criteria: Individual participant data can be shared if the principal investigator is contacted.

REFERENCES:
- [Result] Linkevicius T, Apse P, Grybauskas S, Puisys A. The influence of soft tissue thickness on crestal bone changes around implants: a 1-year prospective controlled clinical trial. Int J Oral Maxillofac Implants. 2009 Jul-Aug;24(4):712-9. PMID 19885413
- [Result] Puisys A, Linkevicius T. The influence of mucosal tissue thickening on crestal bone stability around bone-level implants. A prospective controlled clinical trial. Clin Oral Implants Res. 2015 Feb;26(2):123-9. doi: 10.1111/clr.12301. Epub 2013 Dec 9. PMID 24313250
- [Result] Linkevicius T, Puisys A, Steigmann M, Vindasiute E, Linkeviciene L. Influence of Vertical Soft Tissue Thickness on Crestal Bone Changes Around Implants with Platform Switching: A Comparative Clinical Study. Clin Implant Dent Relat Res. 2015 Dec;17(6):1228-36. doi: 10.1111/cid.12222. Epub 2014 Mar 28. PMID 24673875
- [Derived] Terzioglu B, Ayyildiz BG. Effect of supracrestal tissue height on marginal bone level changes at platform-switching dental implants placed crestally and subcrestally: A randomized clinical-trial. J Dent. 2024 Sep;148:105219. doi: 10.1016/j.jdent.2024.105219. Epub 2024 Jul 1. PMID 38960001